CLINICAL TRIAL: NCT05680155
Title: A Phase 3, Multi-center, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of XW003 in Patients With T2DM Inadequately Controlled by Diet and Exercise Alone
Brief Title: A Phase 3 Study to Evaluate the Efficacy of XW003 Compared With Placebo in T2DM Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW0502-1031
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2023-07

CONDITIONS: T2DM; Type 2 Diabetes Mellitus
Keywords: T2DM; Glucagon-like peptide-1; Ecnoglutide; XW003; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- C1-XW003 (Experimental): High dosage of XW003 once weekly
  Interventions: Drug: Ecnoglutide
- C1-Placebo (Placebo Comparator): Matched Placebo once weekly
  Interventions: Drug: Placebo
- C2-XW003 (Experimental): Low dosage of XW003 once weekly
  Interventions: Drug: Ecnoglutide
- C2-Placebo (Placebo Comparator): Matched Placebo once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecnoglutide — Subcutaneous Injection
  Other Names: XW003
  Arms: C1-XW003; C2-XW003
Drug: Placebo — Subcutaneous Injection with matched volume
  Arms: C1-Placebo; C2-Placebo

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of XW003 versus placebo in patients with type 2 diabetes mellitus (T2DM) inadequately controlled by diet and exercise alone

DETAILED DESCRIPTION:
In this Phase 3 study, eligible participants will be randomized in a 2:2:1:1 ratio to receive once-weekly subcutaneous XW003 (high or low dose) or volume matching placebo as an adjunct to lifestyle intervention for 24 weeks. The core treatment phase will be followed by a 28-week open-label period where all participants receive XW003.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to participate in the study, give written informed consent, and comply with the study specific requirements and all protocol procedures.
2. Sex: male or female; Age: 18 to 75 years, inclusive
3. BMI: 20.0 kg/m^2 to 35.0 kg/m^2, inclusive
4. Have been diagnosed with T2DMthat is inadequately controlled with at least 3 months of diet and exercise prior to screening.
5. HbA1c ranging from 7.5% to 11.0% at screening, inclusive
6. FPG ≤13.9 mmol/L at screening.

Exclusion Criteria:

1. History of type 1 or other types of diabetes mellitus.
2. Use of any GLP-1 analogue during the 3 months preceding to screening.
3. History of proliferative diabetic retinopathy, diabetic maculopathy, diabetic neuropathy, or diabetic foot during the 6 months preceding screening.
4. History of acute or chronic pancreatitis or high risk factors for pancreatitis.
5. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
6. History of stomach surgeries or disorders associated with slowed emptying of the stomach during the past 6 months.
7. History of heart attack, stroke, or congestive heart failure of Grade 3 or 4 in the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, Week 24

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline, Week 5, Week 9, Week 13, Week 17, Week 29, Week 33, Week 37, Week 45, Week 52
Proportion of subjects with HbA1c < 7% and HbA1c ≤6.5% after treatment | week 24, week 52
Proportion of subjects with HbA1c < 7%, with no severe hypoglycemia or no weight gain | week 24
Change from baseline in fasting plasma glucose (FPG) | Baseline, Week 24 and Week 52
Change from baseline in fasting insulin | Baseline, Week 24 and Week 52
Change from baseline in lipid panel | Baseline, Week 24 and Week 52
Change from baseline in 2-hour postprandial blood glucose | Baseline, Week 24 and Week 52
Change from baseline in 7-point self-monitored blood glucose | Baseline, Week 24 and Week 52
Change from baseline in HOMA-IR | Baseline, Week 24 and Week 52
Change from baseline in HOMA-β | Baseline, Week 24 and Week 52
Change from baseline in body weight | Baseline, Week 24 and Week 52
Change from baseline in waist circumference | Baseline, Week 24 and Week 52
Change from baseline in hip circumference | Baseline, Week 24 and Week 52

OTHER OUTCOMES:
Incidence of adverse events | from baseline to EOS
Pharmacokinetics: plasma trough level of XW003 | Baseline, D29, D57, D85, D168, D197, D225, D253, D364, D399
Immunogenecity of XW003 | Baseline, D85, D168, D253, D399

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu D, Wang W, Tong G, Ma J, Wen B, Zheng X, Shi B, Pang S, Wang K, Shi X, Zhang X, Fu L, Liu Y, Lu Y, Huang D, Jiang C, Pan T, Xue H, Han J, Ding H, Bing S, Jiang F, Zheng Q, Yang M, Guan L, Liu X, Ning J, Bu Y, Guo M, Yang L, Guo W, Li Y, Xu S, Pan H. Efficacy and safety of cAMP signalling-biased GLP-1 analogue ecnoglutide monotherapy versus placebo in patients with type 2 diabetes (EECOH-1): a multi-centre, randomised, double-blind, placebo-controlled, phase 3 trial. Nat Commun. 2026 Jan 7;17(1):1420. doi: 10.1038/s41467-025-68165-7. PMID 41501026